CLINICAL TRIAL: NCT03775304
Title: Evaluation of the Relevance Indicators of Quality of Care for Dying Patients Based on Analysis of Care and Follow-up Course of the Leonetti Law. EFIQUAVIE Study
Brief Title: Evaluation of End of Life Quality of Care
Acronym: EFIQUAVIE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI10031
Record Dates: First submitted 2018-12-06; First posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2017-03

CONDITIONS: Neoplasm Malignant; Quality of Life; End of Life Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study uses a mixed method study to evaluate wether the use of the indicators of the Quality of end-of-life cancer care, developed by Earle et al [Earle JCO 2003; DOI: 10.1200/JCO.2003.03.059] would be relevant and measurable in France. The qualitative part of study was designed to investigate the representations of quality by face-to face interviews with family carer of recently deceased cancer patients, and with their oncologists, and nurses. The quantitative part of the study, consisted in a decedents case series analysis, diagnosed with advanced cancer and followed up in 5 centers. Data on trajectory of care were collected from different complementary sources associating national mortality data, hospital activity data, and health records.

The study was approved by the French data protection authority (CNIL) number 611273.

ELIGIBILITY:
Inclusion criteria

* Patients aged ≥ 18,
* diagnosed with advanced cancer (recruited from hospital activity data, by a stay with a ICD code of metastatic cancer between Oct 1st, 2009 and Dec 31, 2010)
* deceased between, Jan 1st, 2010 and Dec 31, 2010 (vital status identified either from hospital activity data, or from national mortality statistics)

Exclusion Criteria:

* diagnosis with non solid tumor (haematology)
* age < 18

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients deceased in 2010, among all patients identified in the DRG database of the 5 participating center with a diagnosis of metastatic cancer, during at least one stay between Oct 1st, 2009 and Dec 31, 2010.
  200 patients per study center were randomly selected for the study.
Sampling Method: Probability Sample
Enrollment: 997 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-15 (Actual)

PRIMARY OUTCOMES:
Use of emergency services within last 30 days before death | Through study completion, up to 1 year

SECONDARY OUTCOMES:
Patients received chemotherapy in the last 14 days of life | Through study completion, up to 1 year
Location of death | Through study completion, up to 1 year
Among patients who died in palliative care unit, those who died within 3 days after admission | Through study completion, up to 1 year
Admission in intensive care unit within last 30 days before death | Through study completion, up to 1 year
Among patients with pain relief opioid treatment, those with combined short term and long acting opioid orders | Through study completion, up to 1 year

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - APHP Hôpital Cochin, Paris
  - APHP Hôpital Européen Georges Pompidou, Paris
  - APHP Hôpital Henri Mondor, Paris
  - Institut Gustave Roussy, Villejuif
  - Institut Curie, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No